CLINICAL TRIAL: NCT05955352
Title: The Effect of Using Perineal Warm Compress Techniques During the Second Stage of Labor on Perineal Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tribhuvan University, Nepal (Other)
Responsible Party: Principal Investigator, Isabel Lawot, Lecturer, Tribhuvan University, Nepal
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TribhuvaU
Record Dates: First submitted 2023-06-21; First posted 2023-07-21 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Heat Therapy; Perineal Tear; Pain; Labor
Keywords: perineal warm compression, Tear, Pain
MeSH Terms: conditions — Hyperthermia; Pain; Lacerations

STUDY DESIGN:
Intervention Model Description: there are two groups randomly selected. intervention and control group, One group will be used perineal heat application and the control group will be received standardized care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Procedural intervention and Control group with standard care (Experimental): There will be two groups. Interventional group will receive perineal warm compression and control group will receive standard care
  Interventions: Procedure: Perineal warm compression Technique

INTERVENTIONS:
Procedure: Perineal warm compression Technique — There will be two groups. Interventional group will receive perineal warm compression and control group will receive standard care to asses the pain intensity and perineal tear
  Other Names: Perineal heat therapy

SUMMARY:
The goal of the clinical trial is to determine the effect of second-stage warm compress application on perineal pain and trauma among primiparous women. The main questions may reveal the pain intensity and the perineal outcome of the warm compress which might be helpful to the women during labor and related authority of the hospital.

The intervention with warm perineal compression will be done among primiparous mothes during second stage of labor

DETAILED DESCRIPTION:
Participants

* After full dilatation of the cervix, assign participants in a 1:1 ratio to the study and control groups randomly.
* Ask women to select one closed envelope containing a card with the group allocation (study or control groups)
* Provide usual care according to the unit protocol to all the women until the second stage of labor.
* Provide the participants of the study group with a warm perineal compress during the whole second stage of labor
* Provide usual care according to the unit protocol to the participants of control group during the whole second stage of labor.

The process of applying the warm perineal compress

* Fill a clean container with warm water (45-59°C)
* Soak a clean pad in the water, squeeze then place gently on the perineum during each uterine contraction.
* Maintain the temperature between 38-44°C during its application.
* Re-soak the pad in warm water between contractions, to maintain warmth and then reapply.
* Replace the water in the container every 15 minutes until delivery or if the temperature drop below 45°C

ELIGIBILITY:
Inclusion Criteria: Low-risk pregnant mothers such as no hypertension, Headache, Bleeding Infection etc -

Exclusion Criteria: Pregnancy with any health problems such as Preeclampsia, Bleeding, Obstructed Labour, Cesarean section

-

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only Female
Enrollment: 46 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
level of pain intensity | 15 minutes after application of warm compression
  Pain intensity will be assessed using an NPRS after the application of warm compression on perineum during the second stage of labor and The scale ranges from 0 to 10, where 0 indicates no pain, and 10 represents the worst level of pain. In between these two extremes, words such as mild, moderate, severe, and very severe pain are assigned to each 2 cm distance on the line, respectively.
Perineal outcomes | 1 hour after application of warm compression
  Perineal outcomes will be assessed as the degree of tears during childbirth as an effect of perineal warm compression

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Lawot, MN, Principal Investigator — Maharajgunj Nursing Campus, Tribhuvan University
Locations (1):
- Tribhuvan University Teaching Hospital, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No